CLINICAL TRIAL: NCT00250965
Title: Magnesium for the Prevention of Atrial Arrhythmias After Cardiac Surgery
Brief Title: MPAACS: Magnesium for the Prevention of Atrial Arrhythmias After Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by DSMB; futility analysis showing Mg treatment not efficacious
Sponsor: University of British Columbia (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Dr. Karin Humphries, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20R20015
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: intravenous magnesium — Subjects will be randomized prior to surgery (1:1) to receive 5 g magnesium or placebo (saline) bolus by the anaesthesiologist upon removal of the crossclamp. On postoperative days 1 through 4, subjects will receive either IV MgSO4 (5g in 250 ml normal saline) or IV placebo (250 ml normal saline) infusion over 4 hours daily.

SUMMARY:
The objective of our research is to determine whether treatment with magnesium will reduce the incidence of atrial fibrillation in patients undergoing cardiac surgery. Several small studies of magnesium have already been conducted, but these studies were small and the results conflicting. A large, well-conducted study of magnesium treatment is required to definitively determine whether magnesium is effective in preventing this common complication after surgery. In addition, our study will include patients undergoing valvular surgery, a group previously excluded from research despite the fact that they are at increased risk of atrial fibrillation.

DETAILED DESCRIPTION:
All patients referred for non-emergent cardiac surgery for isolated CABG, isolated valvular heart surgery, or combined valvular and CABG surgery are eligible for the study. Subjects will be randomized prior to surgery (1:1) to receive 5 g magnesium or placebo (saline) bolus by the anaesthesiologist upon removal of the crossclamp. On postoperative days 1 through 4, subjects will receive either IV MgSO4 (5g in 250 ml normal saline) or IV placebo (250 ml normal saline) infusion over 4 hours daily. Atrial fibrillation (and other arrhythmias) will be detected by placing all subjects on continuous 24-hour ECG telemetry monitoring for postoperative days 0 through 4.

The study is powered to detect at least a 30% relative reduction in postoperative atrial fibrillation in the CABG group; n=756. Because of the higher incidence of atrial fibrillation in the Valve +/- CABG group a total of 500 patients will be required to detect at least a 30% difference between treatment groups. These sample sizes are based on an alpha of 0.05 and 80% power.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing coronary artery bypass surgery with or without valve procedure
* scheduled for on-pump or cardiopulmonary bypass protocol

Exclusion Criteria:

* existing atrial fibrillation/flutter in the past year or on antiarrhythmic medications
* ventricular fibrillation
* sustained ventricular tachycardia
* 2nd or 3rd degree heart block
* paroxysmal supraventricular tachycardia
* major aortic repair planned during open-heart procedure
* permanent atrial/ventricular pacemaker implanted
* dialysis dependent or creatinine clearance < 35 umoles/min or oliguric/anuric renal failure
* patient intolerant of beta blockers
* patient has reactive airways disease dependent on regular beta-adrenergic agents
* patient is scheduled to undergo off-pump surgical protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 927 (Actual)
Dates: Start 2004-07; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation | 0-4 days after surgery

SECONDARY OUTCOMES:
stroke | 0-4 days after surgery
death | 0-4 days after surgery
myocardial infarction | 4 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karin H Humphries, DSc, Principal Investigator — University of British Columbia/St. Paul's Hospital; Hubert Wong, PhD, Study Chair — University of British Columbia, Department of Health Care & Epidemiology
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia